CLINICAL TRIAL: NCT04992546
Title: A Randomized, Intra-patient, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Topically Administered PRN473 (SAR444727) in Patients With Mild to Moderate Atopic Dermatitis
Brief Title: Phase 2a Study of the Safety, Tolerability, and Pharmacokinetics of Topically Administered PRN473 (SAR444727) in Patients With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Principia Biopharma, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT17131; U1111-1260-4204 (Registry Identifier: ICTRP); PRN473-0005 (Other: Principia Biopharma)
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — PRN473

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR444727 5% BID per lesion (Experimental): During the double-blinded period, 2 target lesions per participant (with difference no greater than 1 point in total sign scores [TSS]) were randomized in 1:1 ratio to receive either SAR44727 Gel 5 percent (%) or matching placebo (i.e., each participant was treated with both SAR444727 5% BID and placebo in parallel). During open-label period, participants applied SAR444727 Gel, 5% twice daily (BID) to the all atopic dermatitis (AD)-affected areas, except the scalp, palms, soles and genitals through Days 15 to 42.
  Interventions: Drug: PRN473 (SAR444727)
- Placebo then SAR444727 5% BID per lesion (Placebo Comparator): Multiple topical doses of placebo for 14 days, and PRN473 (SAR444727) for 28 days
  Interventions: Drug: PRN473 (SAR444727); Drug: Placebo

INTERVENTIONS:
Drug: PRN473 (SAR444727) — White to off-white gel suspension
Drug: Placebo — White to off-white gel suspension
  Arms: Placebo then SAR444727 5% BID per lesion

SUMMARY:
This was a Ph2a study that consists of a double-blind, intra-patient placebo-controlled treatment period and an open-label uncontrolled treatment period with objective to evaluate the safety, tolerability, PK and preliminary efficacy of PRN473 in up to 40 patients with mild to moderate AD.

On Day 1 (Baseline) of the Blinded Period, 2 target lesions with a difference no greater than 1 point in Total Sign Score (TSS) were randomly assigned to treatment in an intra-patient 1:1 manner, one lesion to PRN473 and the other to matching placebo.

Participation took approximately 13 weeks, including up to a 5-week screening period, a 6-week treatment period, end of study assessments 1 day after last dose, and a safety follow-up phone call 2 weeks after last dose.

DETAILED DESCRIPTION:
Study duration per patient was approximately 56 days including a 42-days treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults 18 to 70 years of age (inclusive) at the time of informed consent.
* Diagnosed with mild to moderate AD.
* History of AD for at least 6 months as determined by the Investigator through patient interview.
* Stable disease for the 4 weeks prior to the screening visit with no significant flares in AD as determined by the Investigator.
* Validated Investigator Global Assessment-atopic dermatitis (vIGA-AD) score of Moderate or Mild at Screening. The vIGA-AD was evaluated for the entire body except scalp, palms, soles and genitals.
* HadAD involvement (excluding scalp, palms, soles and genitals) of at least 1.0% BSA and no more than 14.0% BSA.
* Had at least two target lesions 100 cm2 or greater with a difference no greater than 1 point in lesion TSS and at least 5 cm apart located on the trunk (excluding genitals) or upper extremities (excluding palms).
* If female, patients with child-bearing potential must have a negative pregnancy test, and agree to practice true abstinence or agree to use highly effective contraception.
* If male, agree to use a male condom and highly effective contraception with female partners of child-bearing potential.
* In good health as judged by the Investigator.

Exclusion Criteria:

* Patients who had failed 2 or more prior systemic treatments for AD.
* Patients who had received a live or attenuated vaccine in the last 12 weeks or intend to receive a live or attenuated vaccine during the study.
* Patients who cannot discontinue prohibited medications and treatments prior to the Baseline visit and during the study.
* Has unstable AD, based on the judgement of the Investigator, or any consistent requirement for high potency topical steroids to manage AD signs or symptoms.
* Patients who had significant active systemic or localized bacterial, viral, fungal, and helminth infection in the last 30 days.
* Patients unwilling to refrain from prolonged sun exposure or use of a tanning bed or other artificial light emitting devices for 4 weeks prior to Baseline and during the study.
* Patients with other skin conditions that would interfere with evaluations of the effect of the study medication on AD, as determined by the Investigator.
* Patients with known genetic dermatological conditions that overlap with AD, such as Netherton syndrome.
* Previous used of a BTK inhibitor.
* Women who were pregnant, wishing to become pregnant during the study, or were breastfeeding.
* Patients were undergoing allergy (eg, food allergy testing or skin prick testing), patch testing, or food challenges, or plan to do so during the study.
* Patients who had undergone major surgery within 4 weeks prior to Day 1 or patients who had a major surgery planned during the study.
* Regular use of drugs of abuse or regular alcohol consumption within 6 months prior to the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (9):
  - Collaborative Neuroscience Research-Site Number:8400004, Long Beach, California
  - California Allergy & Asthma Medical Group-Site Number:8400008, Los Angeles, California
  - Florida International Research Center-Site Number:8400017, Miami, Florida
  - Lenus Research & Medical Group-Site Number:8400006, Sweetwater, Florida
  - Clinical Research Trials of Florida, Inc-Site Number:8400013, Tampa, Florida
  - Remington Davis Inc-Site Number:8400012, Columbus, Ohio
  - J&S Studies-Site Number:8400015, Bryan, Texas
  - Center for Clinical Studies, LTD. LLP-Site Number:8400014, Houston, Texas
  - Progressive Clinical Research-Site Number:8400002, San Antonio, Texas
- Canada (3):
  - Investigational Site Number :1240008, Hamilton, Ontario
  - Investigational Site Number :1240007, London, Ontario
  - Investigational Site Number :1240002, Québec

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT17131 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25209&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 12 centers in 2 countries. A total of 74 participants were screened from 13 Aug 2021 to 27 Oct 2022, of which 35 were screen failures due to not meeting eligibility criteria.
Pre-assignment Details: A total of 39 participants were randomized during the double-blind period and a total of 38 participants entered the open-label period. The study included a 5-week screening period, a 6-week treatment period that included double blinded-period from Days 1 to 14 and an open-label period from Days 15 to 42, end of study/early termination Day 43, and a safety follow-up 2 weeks after the last dose.
Units Other Than Participants: lession
Groups:
- SAR444727 5% BID+Placebo (Double Blinded Period), Then SAR444727 5% BID (Open Label Period): During the double-blinded period, 2 target lesions per participant (with difference no greater than 1 point in total sign scores [TSS]) were randomized in 1:1 ratio to receive either SAR44727 Gel 5 percent (%) or matching placebo in parallel (i.e., each participant was treated with both SAR444727 5% BID and placebo). During open-label period, participants applied SAR444727 Gel, 5% twice daily (BID) to the all atopic dermatitis (AD)-affected areas, except the scalp, palms, soles and genitals through Days 15 to 42.
Period: Double-Blinded Treatment Period
Arm/Group | SAR444727 5% BID+Placebo (Double Blinded Period), Then SAR444727 5% BID (Open Label Period)
Started | 39; 78 lession
Completed | 37; 74 lession
Not Completed | 2; 4 lession
Not completed — Withdrawal by Subject | 1
Not completed — Doses missed due to Covid-19 pandemic circumstances at the site | 1
Period: Open-Label Treatment Period
Arm/Group | SAR444727 5% BID+Placebo (Double Blinded Period), Then SAR444727 5% BID (Open Label Period)
Started | 38; 76 lession (One participant discontinued due to Covid at Day 12 and re-entered Open-label treatment period after Covid recovery.)
Completed | 34; 68 lession
Not Completed | 4; 8 lession
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The randomized population included all participants from the screened population who had been allocated to a randomized treatment by interactive response technology (IRT) regardless of whether the treatment was received.
Groups:
- SAR444727 5% BID+Placebo (Double-blinded Period), Then SAR444727 5% BID (Open Label Period): During the double-blinded period, 2 target lesions per participant (with difference no greater than 1 point in total sign scores [TSS]) were randomized in 1:1 ratio to receive either SAR44727 Gel 5 percent (%) or matching placebo in parallel (i.e., each participant was treated with both SAR444727 5% BID and placebo). During open-label period, participants applied SAR444727 Gel, 5% twice daily (BID) to the all atopic dermatitis (AD)-affected areas, except the scalp, palms, soles and genitals through Days 15 to 42.
Arm/Group | SAR444727 5% BID+Placebo (Double-blinded Period), Then SAR444727 5% BID (Open Label Period)
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 12
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP. SAEs were any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were AEs that occurred from the time of the first IMP in the safety analysis period.
Time Frame: From the first IMP administration (Day 1) up to Day 58
Population: The Safety population included all randomized participants who received any amount of IMP. TEAE and TESAE were assessed per patient according to study design.
Measure: Count of Participants; unit: Participants
Groups:
- SAR444727 5% BID+Placebo: Double Blinded Period: During the double-blinded period, 2 target lesions per participant (with difference no greater than 1 point in TSS) were randomized in 1:1 ratio to receive either SAR44727 Gel 5% or matching placebo (i.e., each participant was treated with both SAR444727 5% BID and placebo in parallel). This group represents the AE which occurred while participants were treated with both SAR444727 5% BID and placebo at the same time.
- SAR444727 5% BID: Open Label Period: During open-label period, participants applied SAR444727 Gel, 5% BID to the all AD-affected areas, except the scalp, palms, soles and genitals through Days 15 to 42.
Arm/Group | SAR444727 5% BID+Placebo: Double Blinded Period | SAR444727 5% BID: Open Label Period
Number analyzed (Participants) | 39 | 38
Participants
  TEAEs | 7 | 12
  TESAEs | 0 | 0

2. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities (PCSA): Vital Signs
Description: Vital signs assessments included supine systolic blood pressure, supine diastolic blood pressure, supine heart rate (HR), and body temperature. Criteria for PCSA: Supine SBP: ≤ 95 mmHg and decrease from baseline ≥ 20 mmHg, ≥ 160 mmHg and increase from baseline ≥ 20 mmHg; Supine DBP : ≤ 45 mmHg and decrease from baseline ≥ 10 mmHg, ≥ 110 mmHg and increase from baseline ≥ 10 mmHg; Orthostatic SBP: ≤ -20 mmHg; Orthostatic DBP: ≤ -10 mmHg; Supine PR: ≤ 50 beats/min and decrease from baseline ≥ 20 beats/min, ≥ 120 beats/min and increase from baseline ≥ 20 beats/min; Weight :≥ 5% decrease from baseline, ≥ 5% increase from baseline
Time Frame: From the first IMP administration (Day 1) up to Day 45
Population: The Safety population included all randomized participants who received any amount of IMP. Only data from the participants analyzed were reported. PCSAs were assessed per patient according to study design.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR444727 5% BID+Placebo (Double Blinded Period), Then SAR444727 5% BID (Open Label Period)
Number analyzed (Participants) | 38
Participants
  Supine systolic blood pressure | 0
  Supine diastolic blood pressure | 0
  Supine HR | 0
  Body temperature | 0

3. Primary Outcome: Number of Participants With PCSA in 12-Lead Electrocardiogram (ECG)
Description: Criteria for PCSA: HR: less than (<) 50 beats per minute (bpm), > 90 bpm, > 90 bpm and increase from baseline > = 20 bpm, > 100 bpm; PR interval: > 200 milliseconds (msec), > 200 msec and increase from baseline >= 25 %, > 220 msec; QRS interval: greater than (>) 110 msec, > 110 msec and increase from baseline greater than or equal to (>=) 25%, > 120 msec; QT interval: > 500 msec; QTc interval > 450 msec; > 480 msec, increase from baseline (30-60) msec, increase from baseline > 60 msec.
Time Frame: From the first IMP administration (Day 1) up to Day 45
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- SAR444727 5% BID+Placebo (Double Blinded Period), Then SAR444727 5% BID (Open Label Period): During the double-blinded period, 2 target lesions per participant (with difference no greater than 1 point in TSS) were randomized in 1:1 ratio to receive either SAR44727 Gel 5% or matching placebo in parallel (i.e., each participant was treated with both SAR444727 5% BID and placebo). During open-label period, participants applied SAR444727 Gel, 5% BID to the all AD-affected areas, except the scalp, palms, soles and genitals through Days 15 to 42.
Arm/Group | SAR444727 5% BID+Placebo (Double Blinded Period), Then SAR444727 5% BID (Open Label Period)
Number analyzed (Participants) | 38
Participants
  HR < 50 bpm | 0
  HR > 90 bpm | 1
  HR > 90 bpm and increase from baseline >= 20 bpm | 0
  HR > 100 bpm | 0
  PR interval > 200 msec | 1
  PR interval > 200 msec and increase from baseline >= 25% | 0
  PR interval > 220 msec | 0
  QRS interval > 110 msec | 2
  QRS interval > 110 msec and increase from baseline >= 25% | 0
  QRS interval > 120 msec | 0
  QT interval > 500 msec | 0
  QTc interval > 450 msec | 1
  QTc interval > 480 msec | 0
  QTc interval increase from baseline (30-60) msec | 2
  QTc interval increase from baseline > 60 msec | 0

4. Primary Outcome: Number of Participants With PCSA: Hematology
Description: Criteria for PCSA: Hemoglobin (Hb) <=115 grams per liter (g/L) (Male[M]) or <=95 g/L (Female[F]), >= 185 g/L (M) or >=165 g/L (F), decrease from baseline >= 20 g/L; Hematocrit: <=0.37 volume/volume (v/v) (M) or <=0.32 v/v (F), >=0.55 v/v (M) or >=0.5 v/v (F); Red blood cells (RBC): >=6 Tera/L; Platelets: < 100 Giga/L, >=700 Giga/L; Neutrophils: <1.5 Giga/L (Non-Black [NB]) or <1.0 Giga/L (Black [B]); Lymphocytes: > 4.0 Giga/L; Monocytes: >0.7 Giga/L; Basophils: >0.1 Giga/L; Eosinophils: >0.5 Giga/L or >upper limit of normal (ULN) (if ULN >=0.5 Giga/L).
Time Frame: From the first IMP administration (Day 1) up to Day 45
Population: The Safety population included all randomized participants who received any amount of IMP. Only those participants with data available were analyzed. PCSAs were assessed per patient according to study design.
Measure: Count of Participants; unit: Participants
Groups:
- SAR444727 5% BID+Placebo: Double Blinded Period: During the double-blinded period, 2 target lesions per participant (with difference no greater than 1 point in TSS) were randomized in 1:1 ratio to receive either SAR44727 Gel 5% or matching placebo (i.e., each participant was treated with both SAR444727 5% BID and placebo in parallel). This group represents the PCSA which occurred while participants were treated with both SAR444727 5% BID and placebo at the same time.
Arm/Group | SAR444727 5% BID+Placebo: Double Blinded Period | SAR444727 5% BID: Open Label Period
Number analyzed (Participants) | 24 | 38
Participants
  Hb <= 115 g/L (M); <= 95 g/L (F) | 0 | 1
  Hb >=185 g/L (M) or >=165 g/L (F) | 0 | 0
  Hb decrease from baseline >=20 g/L | 0 | 0
  Hematocrit <=0.37 v/v (M) or <=0.32 v/v (F) | 0 | 1
  Hematocrit >=0.55 v/v (M) or >=0.5 v/v (F) | 0 | 0
  RBC >=6 Tera/L | 0 | 0
  Platelets <100 Giga/L | 0 | 0
  Platelets >=700 Giga/L | 0 | 0
  Neutrophils <1.5 Giga/L (NB) or <1.0 Giga/L (B) | 0 | 0
  Lymphocytes: > 4.0 Giga/L | 1 | 2
  Monocytes: >0.7 Giga/L | 2 | 7
  Basophils: >0.1 Giga/L: number analyzed (Participants) | 0 | 0
  Eosinophils: >0.5 Giga/L or > ULN (ULN >=0.5 Giga/L): number analyzed (Participants) | 0 | 0

5. Primary Outcome: Number of Participants With PCSA: Electrolyte Parameters
Description: Criteria for PCSA: Sodium: <=129 millimoles (mmol)/L, >=160 mmol/L; Potassium: <3 mmol/L, >=5.5 mmol/L and Chloride: <80 mmol/L, >115 mmol/L.
Time Frame: From the first IMP administration (Day 1) up to Day 45
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | SAR444727 5% BID+Placebo: Double Blinded Period | SAR444727 5% BID: Open Label Period
Number analyzed (Participants) | 24 | 38
Participants
  Sodium <=129 mmol/L | 0 | 0
  Sodium >=160 mmol/L | 0 | 0
  Potassium <3 mmol/L | 0 | 0
  Potassium >=5.5 mmol/L | 1 | 1
  Chloride <80 mmol/L | 0 | 0
  Chloride >115 mmol/L | 0 | 0

6. Primary Outcome: Number of Participants With PCSA: Metabolic Parameters
Description: Criteria for PCSA: Glucose: <=3.9 mmol/L and < lower limit of normal range (LLN); >=11.1 mmol/L (unfasted [unfas]) or >=7 mmol/L (fasted [fas]); Albumin: <=25 g/L; Creatine kinase (CK): > 3 ULN, > 10 ULN; C-Reactive protein: > 2 ULN or 10 mg(milligram)/L (if ULN not provided).
Time Frame: From the first IMP administration (Day 1) up to Day 45
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- SAR444727 5% BID+Placebo: Double Blinded Period: During the double-blinded period, 2 target lesions per participant (with difference no greater than 1 point in total sign scores [TSS]) were randomized in 1:1 ratio to receive either SAR44727 Gel 5 percent (%) or matching placebo (i.e., each participant was treated with both SAR444727 5% BID and placebo in parallel). This group represents the PCSA which occurred while participants were treated with both SAR444727 5% BID and placebo at the same time.
Arm/Group | SAR444727 5% BID+Placebo: Double Blinded Period | SAR444727 5% BID: Open Label Period
Number analyzed (Participants) | 24 | 38
Participants
  Glucose <=3.9 mmol/L and <LLN | 0 | 0
  Glucose >=11.1 mmol/L (unfas) or >=7 mmol/L (fas) | 2 | 4
  Albumin <=25 g/L | 0 | 0
  CK > 3 ULN | 1 | 0
  CK > 10 ULN | 1 | 0
  C-Reactive protein: > 2 ULN or 10 mg/L (if ULN not provided): number analyzed (Participants) | 23 | 38
  C-Reactive protein: > 2 ULN or 10 mg/L (if ULN not provided) | 1 | 5

7. Primary Outcome: Number of Participants With PCSA: Renal Function Parameters
Description: Criteria for PCSA: Creatinine: >=150 micromoles per liter (mcmol/L), >=30% change from baseline, >=100% change from baseline.
Time Frame: From the first IMP administration (Day 1) up to Day 45
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | SAR444727 5% BID+Placebo: Double Blinded Period | SAR444727 5% BID: Open Label Period
Number analyzed (Participants) | 24 | 38
Participants
  Creatinine >=150 mcmol/L | 0 | 0
  Creatinine >=30% change from baseline | 1 | 3
  Creatinine >=100% change from baseline | 0 | 0

8. Primary Outcome: Number of Participants With PCSA: Liver Function Parameters
Description: Liver function parameters assessments included alanine transaminase (ALT), aspartate transaminase (AST), alkaline phosphatase, lactate dehydrogenase, total bilirubin, direct bilirubin, and gamma glutamyl transferase (GGT).
Time Frame: From the first IMP administration (Day 1) up to Day 45
Population: The Safety population included all randomized participants who received any amount of IMP. PCSAs were assessed per patient according to study design.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR444727 5% BID+Placebo: Double Blinded Period | SAR444727 5% BID: Open Label Period
Number analyzed (Participants) | 39 | 38
Participants
  ALT | 0 | 0
  AST | 0 | 0
  Alkaline phosphatase | 0 | 0
  Lactate dehydrogenase | 0 | 0
  Total bilirubin | 0 | 0
  Direct bilirubin | 0 | 0
  GGT | 0 | 0

9. Primary Outcome: Number of Participants With PCSA: Urinalysis
Description: Urinalysis parameters assessments included potential of Hydrogen (pH), urobilinogen, and specific gravity.
Time Frame: From the first IMP administration (Day 1) up to Day 45
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SAR444727 5% BID+Placebo: Double Blinded Period | SAR444727 5% BID: Open Label Period
Number analyzed (Participants) | 39 | 38
Participants
  pH | 0 | 0
  Urobilinogen | 0 | 0
  Specific gravity | 0 | 0

10. Primary Outcome: Percentage of Participants With Application-Site Event During Double-Blind Period
Description: Grading of application-site local tolerability symptoms (burning, pruritus, and erythema) were recorded using the grading scale following each dosing during the double-blind period. Grading of application site tolerability symptoms graded from 0 (none) to 3 (severe).
Time Frame: From the first IMP administration (Day 1) up to Week 2
Population: The Safety population included all randomized participants who received any amount of IMP.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Double Blinded Period: During the double blinded period, 2 target lesions per participant (with difference no greater than 1 point in TSS) were randomized in 1:1 ratio to receive either SAR44727 Gel 5% or matching placebo.
- SAR444727 5% BID: Double Blinded Period: During double blinded period, participants applied SAR444727 Gel, 5% BID to the all AD-affected areas, except the scalp, palms, soles and genitals through Days 15 to 42.
Arm/Group | Placebo: Double Blinded Period | SAR444727 5% BID: Double Blinded Period
Number analyzed (Participants) | 38 | 39
percentage of participants
  Burning | 23.7 | 17.9
  Pruritus | 31.6 | 25.6
  Erythema | 47.4 | 48.7

11. Secondary Outcome: Maximum Plasma Concentration (Cmax) of SAR444727
Description: Plasma samples were collected at indicated timepoints for assessment of SAR444727 concentrations.
Time Frame: Day 1, 4 hours post-dose; Day 15, 1 hour post-dose and Day 43, 12 hours post-dose
Population: The Pharmacokinetic (PK) population included all participants who received any amount of IMP and had at least 1 PK sample. Only those participants with data available were analyzed.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | SAR444727 5% BID+Placebo (Double-blinded Period), Then SAR444727 5% BID (Open Label Period)
Number analyzed (Participants) | 36
nanogram/milliliter
  Day 1, 4 hours post-dose | 0 (0.096)
  Day 15, 1 hour post-dose: number analyzed (Participants) | 31
  Day 15, 1 hour post-dose | 0 (0.152)
  Day 43, 12 hours post-dose: number analyzed (Participants) | 35
  Day 43, 12 hours post-dose | 0 (0.035)

ADVERSE EVENTS:
Time Frame: TEAE data was collected from the first IMP administration (Day 1) up to Day 58
Description: Analysis was performed on the safety population. As is pre-specified in the study protocol, all adverse events were collected at the participant level.
Groups:
- SAR444727 5% BID+Placebo: Double Blinded Period: During the double-blinded period, 2 target lesions per participant (with difference no greater than 1 point in total sign scores [TSS]) were randomized in 1:1 ratio to receive either SAR44727 Gel 5 percent (%) or matching placebo (i.e., each participant was treated with both SAR444727 5% BID and placebo in parallel). This group represents the AE which occurred while participants were treated with both SAR444727 5% BID and placebo at the same time.
Arm/Group | SAR444727 5% BID+Placebo: Double Blinded Period | SAR444727 5% BID: Open Label Period
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 7/39 | 12/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAR444727 5% BID+Placebo: Double Blinded Period (N=39) | SAR444727 5% BID: Open Label Period (N=38)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1)
Application site urticaria (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT04992546/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT04992546/SAP_001.pdf